CLINICAL TRIAL: NCT00451984
Title: Hepatitis Vaccination in HIV Infection: Role of Adjuvant Interleukin-2
Acronym: HEPVACHIV
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aalborg University Hospital (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: VN2005/32
Record Dates: First submitted 2007-03-23; First posted 2007-03-26 (Estimated); Last update posted 2007-11-01 (Estimated); Status verified 2007-10

CONDITIONS: HIV Infections; Hepatitis A; Hepatitis B
Keywords: interleukin-2; vaccination; treatment experienced
MeSH Terms: conditions — HIV Infections; Hepatitis A; Hepatitis B | interventions — twinrix; Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: Twinrix
Biological: interleukin-2

SUMMARY:
The response to vaccination for hepatitis is reduced in patients with HIV infection. The hypothesis of the study is that adjuvant interleukin-2 administered subcutaneously at the time of vaccination improves the response rate.

ELIGIBILITY:
Inclusion Criteria:

* Adults with stable antiretroviral therapy and negative for hepatitis A or B

Exclusion Criteria:

* Prior hepatitis A or B

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2007-03

PRIMARY OUTCOMES:
Antibody response to hepatitis A and hepatitis B

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Nielsen, MD, DMSci, Study Chair — Aalborg Hospital, DK-9000 Aalborg, Denmark
Locations (2):
- Denmark (2):
  - Department of Infectious Diseases, Aalborg Hospital, Aalborg
  - Department of Infectious Diseases, Skejby Hospital, Aarhus